CLINICAL TRIAL: NCT01409720
Title: Isometric Muscle Training of the Spine Musculature in Patients With Spinal Bony Metastases Under Radiation Therapy
Brief Title: Isometric Muscle Training in Patients With Spinal Bony Metastases Under Radiation Therapy
Acronym: DISPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. Dr. J. Debus, Dept of Radiation Oncology, University of Heidelberg, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISPO
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2011-08

CONDITIONS: Vertebral Bony Metastases
Keywords: bony metastases; physical exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): patients in arm A carry out daily physical training consisting of three different isometric exercises under the guidance and supervision of a physiotherapist. Training starts day one (first radiotherapy session), 10 daily units of 30 min each are scheduled during radiotherapy. Patients are expected to continue training until 12 weeks post completion of radiotherapy at home.
  Interventions: Other: exercise
- B (No Intervention): Patients in arm B (control group) receive 10 daily sessions of 15 min manual therapy (i.e. massage, etc) starting from day one of radiotherapy.

INTERVENTIONS:
Other: exercise — tailored isometric physical exercise
  Arms: A

SUMMARY:
Standard indications for palliative radiation of bony metastases include pain, spinal cord compression, and impending pathologic fractures.

Palliative radiation therapy serves to reduce pain, improve quality of life, and avoid complications. Tailored training of the paravertebral musculature may support radiation therapy and improve above named factors. DISPO was designed to investigate the impact of tailored physical exercise in patients with vertebral metastases as compared to manual therapy (massage etc.). The trial includes patients with painful bony metastases, patients with spinal cord compression or impending pathological fractures are excluded. The investigations are carried out in a prospective randomized controlled phase-II parallel group design.

DETAILED DESCRIPTION:
Standard indications for palliative radiation of bony metastases include pain, spinal cord compression, and impending pathologic fractures.

Palliative radiation therapy serves to reduce pain, improve quality of life, and avoid complications. Tailored training of the paravertebral musculature may support radiation therapy and improve above named factors. DISPO was designed to investigate the impact of tailored physical exercise in patients with vertebral metastases as compared to manual therapy (massage etc.). The trial includes patients with painful bony metastases, patients with spinal cord compression or impending pathological fractures are excluded. The investigations are carried out in a prospective randomized controlled phase-II parallel group design.

Patients are randomized to one of the following groups: patients in arm A carry out daily physical training consisting of three different isometric exercises under the guidance and supervision of a physiotherapist. Training starts day one (first radiotherapy session), 10 daily units of 30 min each are scheduled during radiotherapy. Patients are expected to continue training until 12 weeks post completion of radiotherapy at home.

Patients in arm B (control group) receive 10 daily sessions of 15 min manual therapy (i.e. massage, etc) starting from day one of radiotherapy.

Follow-up of the patients is scheduled at 12 weeks post completion of radiotherapy incl. CT of the spine and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* solitary or multiple vertebral metastases
* thoracic spine
* lumbar spine
* sacrum
* indication for palliative radiation therapy
* age: 18 - 80 years
* Karnofsky index > 70%
* bisphosphonate therapy inititated

Exclusion Criteria:

* bony metastases of cervical spine or pelvis
* impending fracture
* other serious illnesses or medical conditions: therapy-refractory unstable heart disease, congestive heart failure NYHA °III and °IV; coagulopathies
* Significant neurological or psychiatric condition including dementia or seizures or other serious medical condition prohibiting the patient's participation in the trial by judgement of the investigators
* Legal incapacity or limited legal capacity
* Positive serum/ urine beta-HCG/ pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
feasibility of isometric exercise in vertebral bony metastases | 12 weeks post completion of radiotherapy
  safety and feasibility of isometric exercise in vertebral bony metastases

SECONDARY OUTCOMES:
progression-free survival (PFS) | 2 years post completion of radiotherapy
  PFS is assessed 2 years post completion of radiotherapy
fracture-free survival (FFS) | 2 years post completion of radiotherapy
  FFS is assessed 2 years post completion of radiotherapy
bone density | 12 weeks post completion radiotherapy
  bone density is assessed 12 weeks post completion of radiotherapy using follow-up CT scan of the spine
pain reduction | end of treatment, 12 and 24 weeks post completion of radiotherapy
  pain is evaluated using the VAS pain scale (0-100 points) at completion and 12/ 24 weeks post completion of radiation therapy
Quality of life | 12 and 24 weeks post completion of therapy
  Quality of life is assessed using the EORTC BM22 questionnaire at 12 and 24 weeks post completion of treatment
Fatigue | 12 and 24 weeks post completion of therapy
  Fatigue is assessed using the EORTC FA13 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, MD PhD, Principal Investigator — Heidelberg University
Locations (1):
- Dept of Radiation Oncology, University of Heidelberg, Germany, Heidelberg, Germany, Germany

REFERENCES:
- [Background] ABRAMS HL, SPIRO R, GOLDSTEIN N. Metastases in carcinoma; analysis of 1000 autopsied cases. Cancer. 1950 Jan;3(1):74-85. doi: 10.1002/1097-0142(1950)3:13.0.co;2-7. No abstract available. PMID 15405683
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Berrettoni BA, Carter JR. Mechanisms of cancer metastasis to bone. J Bone Joint Surg Am. 1986 Feb;68(2):308-12. No abstract available. PMID 3753707
- [Background] Bubendorf L, Schopfer A, Wagner U, Sauter G, Moch H, Willi N, Gasser TC, Mihatsch MJ. Metastatic patterns of prostate cancer: an autopsy study of 1,589 patients. Hum Pathol. 2000 May;31(5):578-83. doi: 10.1053/hp.2000.6698. PMID 10836297
- [Background] Cheville AL, Girardi J, Clark MM, Rummans TA, Pittelkow T, Brown P, Hanson J, Atherton P, Johnson ME, Sloan JA, Gamble G. Therapeutic exercise during outpatient radiation therapy for advanced cancer: Feasibility and impact on physical well-being. Am J Phys Med Rehabil. 2010 Aug;89(8):611-9. doi: 10.1097/PHM.0b013e3181d3e782. PMID 20531162
- [Background] Harrington KD. Impending pathologic fractures from metastatic malignancy: evaluation and management. Instr Course Lect. 1986;35:357-81. PMID 3819423
- [Background] Hochschild J. Strukturen und Funktionen begreifen. Funktionelle Anatomie Band 1 und 2, Stuttgart: Thieme
- [Background] Krempien B. Die Entstehung von Knochenschmerzen bei Knochenmetastasen und ihre Behandlung durch Bisphosphonate. Hrsg: Bartsch HH, Hornstein W: Interdisziplinäre Schmerztherapie bei Tumorpatienten, 1998
- [Background] Murnane A, Geary B, Milne D. The exercise programming preferences and activity levels of cancer patients undergoing radiotherapy treatment. Support Care Cancer. 2012 May;20(5):957-62. doi: 10.1007/s00520-011-1167-z. Epub 2011 Apr 27. PMID 21523349
- [Background] Nikander R, Sievanen H, Ojala K, Oivanen T, Kellokumpu-Lehtinen PL, Saarto T. Effect of a vigorous aerobic regimen on physical performance in breast cancer patients - a randomized controlled pilot trial. Acta Oncol. 2007;46(2):181-6. doi: 10.1080/02841860600833145. PMID 17453366
- [Background] Pilge H, Holzapfel BM, Prodinger PM, Hadjamu M, Gollwitzer H, Rechl H. [Diagnostics and therapy of spinal metastases]. Orthopade. 2011 Feb;40(2):185-93; quiz 194-5. doi: 10.1007/s00132-010-1738-6. German. PMID 21271338
- [Background] Roe JW, Ashforth KM. Prophylactic swallowing exercises for patients receiving radiotherapy for head and neck cancer. Curr Opin Otolaryngol Head Neck Surg. 2011 Jun;19(3):144-9. doi: 10.1097/MOO.0b013e3283457616. PMID 21430531
- [Background] Stevinson C, Fox KR. Feasibility of an exercise rehabilitation programme for cancer patients. Eur J Cancer Care (Engl). 2006 Sep;15(4):386-96. doi: 10.1111/j.1365-2354.2006.00677.x. PMID 16968322
- [Background] Verger E, Salamero M, Conill C. Can Karnofsky performance status be transformed to the Eastern Cooperative Oncology Group scoring scale and vice versa? Eur J Cancer. 1992;28A(8-9):1328-30. doi: 10.1016/0959-8049(92)90510-9. PMID 1515244
- [Background] Zhong H, De Marzo AM, Laughner E, Lim M, Hilton DA, Zagzag D, Buechler P, Isaacs WB, Semenza GL, Simons JW. Overexpression of hypoxia-inducible factor 1alpha in common human cancers and their metastases. Cancer Res. 1999 Nov 15;59(22):5830-5. PMID 10582706
- [Derived] Rief H, Bruckner T, Schlampp I, Bostel T, Welzel T, Debus J, Forster R. Resistance training concomitant to radiotherapy of spinal bone metastases - survival and prognostic factors of a randomized trial. Radiat Oncol. 2016 Jul 27;11:97. doi: 10.1186/s13014-016-0675-x. PMID 27464793
- [Derived] Rief H, Omlor G, Akbar M, Bruckner T, Rieken S, Forster R, Schlampp I, Welzel T, Bostel T, Roth HJ, Debus J. Biochemical markers of bone turnover in patients with spinal metastases after resistance training under radiotherapy--a randomized trial. BMC Cancer. 2016 Mar 17;16:231. doi: 10.1186/s12885-016-2278-1. PMID 26983672
- [Derived] Rief H, Petersen LC, Omlor G, Akbar M, Bruckner T, Rieken S, Haefner MF, Schlampp I, Forster R, Debus J, Welzel T; German Bone Research Group. The effect of resistance training during radiotherapy on spinal bone metastases in cancer patients - a randomized trial. Radiother Oncol. 2014 Jul;112(1):133-9. doi: 10.1016/j.radonc.2014.06.008. Epub 2014 Jul 7. PMID 25012645
- [Derived] Rief H, Akbar M, Keller M, Omlor G, Welzel T, Bruckner T, Rieken S, Hafner MF, Schlampp I, Gioules A, Debus J. Quality of life and fatigue of patients with spinal bone metastases under combined treatment with resistance training and radiation therapy- a randomized pilot trial. Radiat Oncol. 2014 Jul 7;9:151. doi: 10.1186/1748-717X-9-151. PMID 24998293
- [Derived] Rief H, Welzel T, Omlor G, Akbar M, Bruckner T, Rieken S, Haefner MF, Schlampp I, Gioules A, Debus J. Pain response of resistance training of the paravertebral musculature under radiotherapy in patients with spinal bone metastases--a randomized trial. BMC Cancer. 2014 Jul 5;14:485. doi: 10.1186/1471-2407-14-485. PMID 24996223
- [Derived] Rief H, Heinhold M, Bruckner T, Schlampp I, Forster R, Welzel T, Bostel T, Debus J, Rieken S; German Bone Research Group. Quality of life, fatigue and local response of patients with unstable spinal bone metastases under radiation therapy--a prospective trial. Radiat Oncol. 2014 Jun 11;9:133. doi: 10.1186/1748-717X-9-133. PMID 24917420
- [Derived] Rief H, Omlor G, Akbar M, Welzel T, Bruckner T, Rieken S, Haefner MF, Schlampp I, Gioules A, Habermehl D, von Nettelbladt F, Debus J. Feasibility of isometric spinal muscle training in patients with bone metastases under radiation therapy - first results of a randomized pilot trial. BMC Cancer. 2014 Feb 5;14:67. doi: 10.1186/1471-2407-14-67. PMID 24499460
- [Derived] Rief H, Jensen AD, Bruckner T, Herfarth K, Debus J. Isometric muscle training of the spine musculature in patients with spinal bony metastases under radiation therapy. BMC Cancer. 2011 Nov 9;11:482. doi: 10.1186/1471-2407-11-482. PMID 22070722